CLINICAL TRIAL: NCT03757858
Title: A Prospective Study of Hyperthermia Combined With Autologous Adoptive Cellular Immunotherapy in the Treatment of Abdominal and Pelvic Malignancies or Metastases
Brief Title: Hyperthermia Combined With Immunotherapy in the Treatment of Abdominal and Pelvic Malignancies or Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director,Capital Medical University (CMU)Cancer Center, Capital Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF8-ACT
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Cancer; Abdominal Cancer; Pelvic Cancer; Metastatic Cancer; Peritoneal Metastases; Liver Metastases
MeSH Terms: conditions — Neoplasms; Pelvic Neoplasms; Neoplasm Metastasis | interventions — Immunotherapy, Adoptive; spartalizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HT+ACT (Experimental)
  Interventions: Device: Thermotron RF-8; Biological: Adoptive cellular Immunotherapy
- HT+ACT+PD-1 (Experimental)
  Interventions: Device: Thermotron RF-8; Biological: Adoptive cellular Immunotherapy; Drug: Anti-PD-1 antibody
- HT+ACT+CT (Experimental)
  Interventions: Device: Thermotron RF-8; Biological: Adoptive cellular Immunotherapy; Drug: Chemotherapy
- HT+CT (Active Comparator)
  Interventions: Device: Thermotron RF-8; Drug: Chemotherapy

INTERVENTIONS:
Device: Thermotron RF-8 — Hyperthermia for 40 minutes, with maximum temperature setted on 42℃ ± 0.5℃ as upper limit, twice a week for a total of 10 times.
Biological: Adoptive cellular Immunotherapy — Mononuclear cells were collected from 50ml peripheral blood , and cultured cytokine-induced killer cells for 15-20 days. Cells were infused back to the patients in 3 times via intravenous infusion .Patients will received at least 2 cycles of CIK Immunotherapy . If the evaluation of the treatment is complete response, partial response or stable disease, additional cycles were eligible.
  Arms: HT+ACT; HT+ACT+CT; HT+ACT+PD-1
Drug: Anti-PD-1 antibody — Patients will receive pembrolizumab 100mg every three weeks and assess the clinical outcome every 2 dosage of anti-PD-1 antibody treatment.
  Arms: HT+ACT+PD-1
Drug: Chemotherapy — Patients will receive standard chemotherapy until disease progression, unacceptable toxicity or patient refusal.
  Arms: HT+ACT+CT; HT+CT

SUMMARY:
It is a non-randomized pilot study.The allocation will be determined by patients or their immediate family members who were cooperative with physician's interpretations on the disease progression and updated information of cutting of edge treatment, the financial affordability, availability of treatment plans, possible tolerance or risks etc.The purpose of this study is to investigate the clinical efficacy and toxicity of autologous cellular immunotherapy combined with hyperthermia in abdominal and pelvic malignancies or metastases patients. Furthermore, to characterize response to different regimens,the investigators intent to explore the predictive and prognostic biomarker, as well as the changes in immune repertoire.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal and pelvic malignancies or metastases
2. Estimated life expectancy > 3 months
3. Age ≥ 18 years old
4. At least one measurable lesion according to the Solid Tumor Evaluation Criteria (RECIST Version 1.1)
5. Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5 (unless patient is receiving warfarin in which case PT-INR must be <3), PTT <1.5X ULN
6. Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.

Exclusion Criteria:

1. Patients with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune related thyroid disease and vitiligo are permitted.
2. Patients with serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
3. Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
4. Concurrent (or within the last 5 years) second malignancy other than non melanoma skin cancer, cervical carcinoma in situ, controlled superficial bladder cancer, or other carcinoma in situ that has been treated.
5. Presence of an active acute or chronic infection including: a urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot). Patients with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
6. Patients on chronic steroid therapy (or other immuno-suppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies or for acute treatment (<5 days) of intercurrent medical condition such as a gout flare) prior to enrollment.
7. Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control while receiving treatment and for a period of 4 months following the last vaccination therapy. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that may be fathered while on this study.
8. Patients with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.
9. There are metal stents or metal fixtures in the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Objective response rate (ORR) | 6 months
  Proportion of patients with reduction in tumor burden of a predefined amount

SECONDARY OUTCOMES:
Progression-free survival of the participants(PFS) | 12 months
  From starting date of the enrollment until the date of first documented disease progression or date of death from any cause, whichever comes first.
Assessment of Patient- Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 12 months
  To assess and compare the PRO-CTCAE by patients in each groups

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical Unvierstiy Cancer Center/ Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided